CLINICAL TRIAL: NCT01480297
Title: A Pilot Study to Determine the Effects of 12 Weeks of Treatment With Salsalate on Measures of Peripheral Neuropathy in Type 1 Diabetes
Brief Title: Pilot Study to Determine Effects of Salsalate in Type 1 Diabetes and Painful Peripheral Neuropathy
Acronym: SALP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Rodica Pop-Busui, Associate Professor of Internal Medicine, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SALP
Record Dates: First submitted 2011-11-23; First posted 2011-11-28 (Estimated); Results first posted 2015-04-24 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Peripheral Neuropathy; Type 1 Diabetes
Keywords: Pain; Neuropathy; Diabetes type 1
MeSH Terms: conditions — Peripheral Nervous System Diseases; Diabetes Mellitus, Type 1; Pain | interventions — salicylsalicylic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Salsalate (Experimental): All subjects will take Salsalate, 3 grams daily (as 3 divided doses of 1 gram with breakfast, lunch and dinner).
  Interventions: Drug: Salsalate

INTERVENTIONS:
Drug: Salsalate — Salsalate 3 grams daily (1 gram TID with meals)
  Other Names: Salsalate (Amneal Pharmaceuticals)

SUMMARY:
This 12 week study will examine the effects of daily Salsalate treatment on markers of neuropathic pain and intra-epidermal nerve fiber density. the study is being done in people with type 1 diabetes with signs and symptoms of peripheral neuropathy.

DETAILED DESCRIPTION:
This project will be used to establish preliminary data for a planned NIH-sponsored multicenter study of the effects of salsalate on diabetic neuropathy (DN) in people with type 1 diabetes. Diabetic peripheral neuropathy (DN) ultimately affects one-half of the patients with type 1 diabetes (T1DM) and is a major cause of disability, high mortality, and poor quality of life. Although intensive glucose control has proven efficacy in delaying or preventing DN in T1DM and type 2 diabetes (T2DM), most people with diabetes do not reach and maintain glycemic levels needed to achieve these benefits. In addition, many patients with diabetes still develop diabetic complications, including DN, despite good glucose control. For DN, no disease modifying treatment other than glycemic control is available. Therefore, it is essential to identify new drug targets and to treat DN as early as possible in its course.

The investigators planned, multi-center study will be the first to determine the effect of an anti-inflammatory agent, salsalate, on DN development and progression, and on DN pain in type 1 diabetes. This proof-of-concept pilot study will measure the effects of short term (12 week) treatment with Salsalate on novel and on established measures of peripheral neuropathy. Ultimately, this may permit measurement of treatment effects over a shorter period of time than by using established measures such as nerve conduction studies. Salsalate, a prodrug form of salicylate, is used to treat osteoarthritis and other rheumatologic conditions. It is highly effective in modulating the IKKβ/NF-κB pathway, with a large margin of safety, and has a glucose lowering effect in patients with type 2 diabetes. The IKKβ/NF-κB pathway is unique in that it is implicated in both the pathogenesis of nerve fiber loss as well as pain in DN. The proposed study design employs a quantifiable early measure of DN, IENFD of the thigh, allowing for accurate assessment of actual nerve fiber density over time.

In the pilot study, biomarkers of pain found in IENF's as well as IENFD will be measured pre and post 3 months of treatment with Salsalate, 3 grams daily.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes (T1D)
* Peripheral neuropathy with symptoms of pain, or with other uncomfortable symptoms (e.g., burning, prickling).
* 18 to 70 years old
* Stable insulin treatment program for at least the past 3 months.
* Abnormal nerve conduction studies (based on study screening examination)
* Willing and able to take an oral (by mouth) medication 3 times per day for 3 months.
* WOMEN using an appropriate method of contraception during the course of the study (hormonal, IUD, or diaphragm.
* Willing and able to provide written informed consent for study participation.

Exclusion Criteria:

* Neuropathy from a cause other than diabetes.
* Allergy to salsalate or similar medications (aspirin, non-steroidal anti-inflammatory medicines like ibuprofen and naproxen).
* Currently on blood thinning agents such as Coumadin, Heparin, Plavix, Pradaxa, high-dose aspirin (more than 325 mg daily).
* Any severe low blood sugar episodes in the past 6 months (needed assistance to treat).
* Diabetic ketoacidosis in the past 6 months.
* Severe neuropathy, or have had an ulcer or amputation on either foot or either leg.
* Creatinine level (a measure of kidney function is greater than 1.4 mg/dl (for women) or greater than 1.5 mg/dl (for men) or your estimated GFR is under 60.
* Albumin in your urine or other signs of reduced kidney function.
* Liver enzymes (including ALT, AST and Bilirubin) levels are more than 2 and ½ times the upper limit of normal.
* Blood platelets are less than 100,000 at the time of screening.
* Organ transplant (lung, kidney, heart, pancreas, liver).
* Chronic immunosuppressive therapy, for example, daily prednisone or other steroids, methotrexate, Imuran, CellCept. This includes daily, or recurrent use of oral steroids used to treat asthma.
* Regular NSAID medications (e.g., Naproxen, Ibuprofen) use. If used occasionally, you will be asked to not use them during the study.
* History of drug or alcohol abuse, or if you take more than 10 alcoholic drinks per week.
* History of stomach ulcers or bleeding from your bowel.
* Heart attack, heart bypass surgery, heart failure or a stroke EVER.
* Current treatment for any cancer (other than basal cell or squamous cell skin cancer).
* Treatment with lithium.
* Ever had Reyes' syndrome.
* Pregnant, nursing, or planning to become pregnant during the time of the study.
* Allergic to lidocaine or epinephrine (used for numbing skin prior to biopsies).
* Keloid scarring in the past.
* Receiving other experimental treatments.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-11; Primary Completion 2012-04 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodica Pop-Busui, MD, PhD, Principal Investigator — University of Michigan, Department of Internal Medicine
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was completed in 3 months time.
Period: Overall Study
Arm/Group | Salsalate
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: adults with type 1 diabetes and painful peripheral neuropathy
Arm/Group | Salsalate
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.0 (5.7)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Intra-epidermal Nerve Fiber Density (IENFD) Fibers Per mm
Description: Intra-epidermal Nerve Fiber Density (IENFD) was measured at two anatomic locations (thigh and ankle) at baseline and after 12 weeks of treatment with Salsalate. IENFD is expressed as fibers per mm. Means and standard deviations are shown.
Time Frame: Baseline and 12 weeks
Population: Type 1 diabetes with painful neuropathy
Measure: Mean (Standard Deviation); unit: fibers per mm
Arm/Group | Salsalate
Number analyzed (Participants) | 8
fibers per mm
  Baseline Thigh IENFD(fibers per mm) | 6.3 (5.4)
  Baseline Ankle IENFD(fibers per mm) | 3.0 (3.3)
  12 Week Thigh IENFD(fibers per mm) | 5.2 (4.4)
  12 Week Ankle IENFD(fibers per mm) | 3.0 (3.5)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Salsalate
Serious Adverse Events (participants affected / at risk) | 1/8
Other Adverse Events (participants affected / at risk) | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Salsalate (N=8)
Severe Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) — Severe hypoglycemia requiring emergency room treatment.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Salsalate (N=8)
Tinnitus (Ear and labyrinth disorders) | 3 (3) — 3 of 8 subjects reported tinnitus. Tinnitus is a known side effect of Salsalate. In all cases, the Tinnitus resolved with decrease in dose, or with cessation of Salsalate treatment.
Upper Respiratory Symptoms (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Cold/Sinusitis
Increased Bleeding from Biopsy Site (Surgical and medical procedures) | 1 (1) — Patient reported increased bleeding from a single biopsy site. Resolved with application of pressure.
Hot Flashes (Endocrine disorders) | 1 (1) — Patient (postmenopausal woman) reported an increase in hot flashes.
Cataract Removal (Eye disorders) | 1 (1) — Scheduled removal of cataracts
Skin Biopsy of Suspicious Lesion (Skin and subcutaneous tissue disorders) | 1 (1) — Patient with suspicious lesion of face - biopsy was benign.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes